CLINICAL TRIAL: NCT00861809
Title: A Multicenter, Double-Blind, Randomized Placebo-Controlled Phase II Study to Evaluate the Pharmacodynamics, Safety, Tolerability, and PK of Single Doses of the Oral Motilin Receptor Agonist GSK962040, in Type 1 Diabetic Male and Female Patients With Gastroparesis
Brief Title: The Effect of Single Doses of the Motilin Receptor Agonist GSK962040 in Type I Diabetic Patients With Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 111809
Record Dates: First submitted 2009-02-26; First posted 2009-03-13 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Gastroparesis
Keywords: single dose; gut motility; Type I Diabetes Mellitus patients; tolerability; phase II; 13C octanoic acid breath test; pharmacodynamics; gastric emtpying; pharmacokinetics
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 Period 1 (Experimental): All patients will receive placebo and 2 of the 3 possible doses of GSK962040 in a randomized, double blind, placebo controlled, incomplete block, three period crossover design.
  Interventions: Drug: GSK962040 25 mg; Drug: Placebo; Drug: GSK962040 50 mg; Drug: GSK962040 1250 mg
- Cohort 1 Period 2 (Experimental): All patients will receive placebo and 2 of the 3 possible doses of GSK962040 in a randomized, double blind, placebo controlled, incomplete block, three period crossover design.
  Interventions: Drug: GSK962040 25 mg; Drug: Placebo; Drug: GSK962040 50 mg; Drug: GSK962040 1250 mg
- Cohort 1 Period 3 (Experimental): All patients will receive placebo and 2 of the 3 possible doses of GSK962040 in a randomized, double blind, placebo controlled, incomplete block, three period crossover design.
  Interventions: Drug: GSK962040 25 mg; Drug: Placebo; Drug: GSK962040 50 mg; Drug: GSK962040 1250 mg

INTERVENTIONS:
Drug: GSK962040 25 mg — 25 mg
Drug: Placebo — placebo comparator
Drug: GSK962040 50 mg — 50 mg
Drug: GSK962040 1250 mg — 125 mg

SUMMARY:
The purpose of this study is to assess the pharmacodynamic effects (gastric emptying), safety, tolerability, and pharmacokinetics of single doses of GSK962040 in Type 1 diabetic patients with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Controlled Type 1 Diabetes Mellitus (glucose < 250 mg/dL) with onset < 30 years of age.
* Male or female between 18 and 70 years of age, inclusive.
* Patient has documented diagnosis of moderate to severe gastroparesis (> 30% at 2 h as determined by scintigraphy; or t1/2b > 109 min as determined by 13C-octanoic acid breath test). All of the following apply:
* Confirmed delayed gastric emptying (properly conducted gastric emptying assessments within last 6 months acceptable) AND a minimum 3 month history of relevant symptoms for gastroparesis (e.g., chronic postprandial fullness, postprandial nausea, vomiting)
* A female patient is eligible to participate if she is of:
* Non-childbearing potential
* Child-bearing potential and agrees to use contraception for at least 4 days following the last dose of study medication.
* Male patients must agree to use contraception from the time of the first dose of study medication through at least 4 days after the last dose of study medication.
* Body weight ≤110 kg and BMI < 32.0 kg/m2 (inclusive).
* Patient has never had a gastrectomy, nor major gastric surgical procedure or any evidence of bowel obstruction within the previous 12 months
* Dosage of any concomitant medications has been stable for at least 3 weeks, except for routine adjustments in daily insulin treatments
* HbA1c level is ≤ 10.0%
* Calculated creatinine clearance > or equal to 50 ml/min
* QTcB or QTcF < 450 msec or QTc<480msec in patients with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Patient has acute severe gastroenteritis
* Patient has a gastric pacemaker
* Patient is on chronic parenteral feeding
* Patient has daily persistent severe vomiting
* Patient has pronounced dehydration
* Patient has had clinical diabetic ketoacidosis in last 4 weeks
* Patient has a history of eating disorders (anorexia nervosa, binge eating, bulimia)
* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study (e.g., prokinetic drugs, macrolide antibiotics (erythromycin))
* Patient is taking opiates.
* Use of prohibited medications listed in Section 9.2 within the restricted timeframe relative to the first dose of study medication.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Presence of thyroid dysfunction (NOTE: patients with abnormal TSH at screening/baseline are not eligible. Patients with a history of hypothyroidism on a stable dose of thyroid replacement therapy are eligible to participate in the study).
* The patient has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test (from the first urine of the day) at screening or prior to dosing.
* Lactating or pregnant females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Patients deemed unable to comply with the procedures outlined in the protocol may be excluded at the Investigator's discretion.
* For male volunteers: An unwillingness of the male patient to comply with the contraception requirements listed in Section 8.1, from the time of the first dose of study medication until at least 4 days following administration of the last dose of study medication.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Gastric emptying, as measured by the 13C octanoic acid breath test (Gastric half emptying time (t1/2b), Duration of the lag time (tlag), Gastric evacuation coefficient (GEC)) | 1.5 h post dose to 5.5 h post dose
Safety and tolerability of GSK962040 (Change from baseline and number of patients outside the normal range for blood pressure, heart rate, 12-lead ECG parameters) | 2 h post dose
Pharmacokinetic parameters of GSK962040: Cmax, Tmax, AUC(0-t), AUC(0-inf) for single-dose, CL/F, V/F, and, if possible, half-life | 24 h post dose
Safety and tolerability of GSK962040 (Adverse events) | 6 weeks
Safety and tolerability of GSK962040 (Change from baseline in clinical chemistry and hematology parameters) | 24 h post dose

SECONDARY OUTCOMES:
Bowel movement parameters (Time to first bowel movement after first dose, Bowel movement count, Stool consistency (Bristol Stool Form scale)) | 24 h post dose
PK/PD relationship of PP, plasma glucagon, GLP-1, and ghrelin after a single dose of GSK962040. | 0-6 h post dose
Plasma glucose | 24 h post dose
Food intake | 24 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Leuven, Belgium
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hellstrom PM, Tack J, Johnson LV, Hacquoil K, Barton ME, Richards DB, Alpers DH, Sanger GJ, Dukes GE. The pharmacodynamics, safety and pharmacokinetics of single doses of the motilin agonist, camicinal, in type 1 diabetes mellitus with slow gastric emptying. Br J Pharmacol. 2016 Jun;173(11):1768-77. doi: 10.1111/bph.13475. Epub 2016 Apr 13. PMID 26924243
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register